CLINICAL TRIAL: NCT03567304
Title: Neurocognitive Function Improvement After Switching From Efavirenz to Rilpivirine in HIV-infected Adults: A Randomized Control Trial
Brief Title: Neurocognitive Function Improvement After Switching From Efavirenz to Rilpivirine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Quanhathai Kaewpoowat, Principal Investigator, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MED-2561-05276
Record Dates: First submitted 2018-06-07; First posted 2018-06-25 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: HIV-1-infection; Neurocognitive Dysfunction
Keywords: HIV; Neurocognitive disorder; Efavirenz; Rilpivirine
MeSH Terms: conditions — Cognition Disorders; Neurocognitive Disorders | interventions — Rilpivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EFV-based (No Intervention): HIV-infected patients, who has been taking efavirenz (EFV)-based regimen for at least 1 year and is diagnosed with asymptomatic neurocognitive impairment (ANI) or mild neurocognitive disease (MND) by neurocognitive battery tests, is randomized to continue EFV-based regimen.
  EFV based regimen defines as efavirenz 600 mg per oral once daily (OD) + 2 Nucleoside Reverse Transcriptase Inhibitors (NRTIs).
- RPV-based (Experimental): HIV-infected patients, who has been taking efavirenz-based regimen for at least 1 year and is diagnosed with asymptomatic neurocognitive impairment (ANI) or mild neurocognitive disease (MND) by neurocognitive battery tests, is randomized to switch antiretroviral therapy to rilpivirine (RPV)-based regimen.
  RPV based regimen defines as rilpivirine 25 mg PO OD + 2 NRTIs.
  Interventions: Drug: Rilpivirine 25 mg

INTERVENTIONS:
Drug: Rilpivirine 25 mg — Rilpivirine 25 mg PO OD with meal (and continue 2 back bone of NRTIs)
  Other Names: Switching from EFV to RPV
  Arms: RPV-based

SUMMARY:
People living with HIV in the era of antiretroviral therapy (ART) continue to suffer high rates of neurocognitive disorder. This is a randomized control trial aiming to evaluate improvement of neurocognitive function after switching efavirenz (EFV) to rilpivirine (RPV). EFV based regimen is currently the first line ART in Thailand. There are several reports suggested that HIV-infected patients who took EFV based regimen had poorer neurocognitive function compared to the comparator. RPV, another first line regimen, has been known to have less neuropsychiatric side effects. We hypothesized that switching EFV to RPV could improve neurocognitive function.

DETAILED DESCRIPTION:
People living with HIV (PLWH) in the era of antiretroviral therapy (ART) continue to suffer high rates of neurocognitive disorder. Previous report revealed that 36% of PLWH in Thailand had this condition. There are several reports suggested that HIV-infected patients who took efavirenz (EFV) based regimen had poorer neurocognitive function compared to the comparator. Rilpivirine (RPV), another first line regimen, has been known to have less neuropsychiatric side effects. We hypothesized that switching EFV to RPV could improve long term neurocognitive function.

PLWH (20 years and older) who received EFV-based regimen for at least 1 years at Chiang Mai University Hospital will be invited to this study. Neurocognitive function will be evaluated using 3 screening questions, International HIV Dementia Scale, Montreal Cognitive Assessment, and comprehensive neurocognitive battery test evaluating 6 different cognitive domains. The participants will be categorized in to 4 groups based on their neurocognitive test results; no evidence of neurocognitive deficit, asymptomatic neurocognitive impairment (ANI), mild neurocognitive disease (MND), and HIV associated dementia (HAD) using Frascati's criteria. The participants with ANI or MND and meet the eligibility criteria will be enrolled to this study. The participants will be randomized in to 2 arms; continuing EFV-based regimen or switching to RPV-based regimen. Neurocognitive function will be evaluated at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection
* Age 20 years old and above
* On EFV-based regimen (EFV and 2 Nucleoside Reverse Transcriptase Inhibitors) for at least 1 year prior to enrollment
* CD4 ≥ 200 cell/mm3 and viral load < 200 copies/mL within 12 months before enrollment
* Able to be read and write in Thai language
* Willing to sign informed consent and able to follow up
* The neurocognitive battery test is compatible with asymptomatic neurocognitive impairment (ANI) or mild neurocognitive disorder (MND) using Frascati's criteria

Exclusion Criteria:

* History of Traumatic Brain Injury, Developmental delay or intellectual deficit, or other neurological conditions have deleterious effects on neurocognitive test based on investigator opinion.
* Active syphilis or on going to treatment with positive for syphilis serological marker (rapid plasma reagin; RPR) in 3 Months before entry study
* Pregnancy
* Renal failure (creatinine clearance < 30 mL/min)
* Transaminitis in the past 3 months (≥5 UNL) Or Decompensated cirrhosis (child-pugh C)
* Moderate depressive score; Patient Health Questionnaire-9 score ≥ 10)
* Positive for any hepatitis B virus and hepatitis C virus serological marker in 3 Months before entry study
* History of treatment failure or drug resistance to EFV and or RPV
* Not suitable or contraindication for RPV (continue proton pump inhibitor drug)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2018-07-06 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Change of neurocognitive function | 12 months
  Improvement is defined by changing neurocognitive status based on Frascati's criteria (using neurocognitive battery tests) 1) from Asymptomatic neurocognitive impairment (ANI) to normal OR 2) from Mild neurocognitive disorder; MND to ANI or normal.

SECONDARY OUTCOMES:
Overall Global Deficit Score of all neurocognitive domains | 12 months
  All neurocognitive domains will be evaluated at 12 months after randomization which include; Verbal and language, Attention and working memory, Abstraction and executive function, Memory (learning, recall), Speed of information processing, and Sensory-perceptual and motor skills. The Global Deficit Score (min of 0, max of 5) of overall performance will be compared.
Adverse reactions after switching from EFV to RPV | 12 months
  Adverse reactions of RPV will be recorded
Prevalence of neurocognitive disorder among HIV-infected patients who has received EFV for at least 1 year | 3 months
  The prevalence of neurocognitive disorder (in percentage), will be evaluated among participants during the screening process.

CONTACTS AND LOCATIONS:
Overall Officials: Quanhathai Kaewpoowat, MD, Principal Investigator — Department of Medicine, Faculty of Medicine, Chiang Mai University, Thailand.
Locations (1):
- Chiang Mai University Hospital, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: Undecided